CLINICAL TRIAL: NCT06979570
Title: Personalized Performance Optimization Platform (P-POP) for Long Duration Spaceflight
Brief Title: Personalized Performance Optimization Platform
Acronym: P-POP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (MIT) (Unknown)
Responsible Party: Principal Investigator, Gary E. Strangman, Principle Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024P003613; 80NSSC21K0669 (Other Grant/Funding Number: National Aeronautics and Space Administration (NASA))
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-05

CONDITIONS: Sensory Science; Performance Assessment; Countermeasure Evaluation; Neurocognitive Function; Psychological Factors
Keywords: Long-Duration Spaceflight; Cogntiive Performance; Wearable Biosensors; Closed-Loop Systems; Auditory Stimulation; Haptic Feedback; Light Modulation; Psychophysiological Monitoring; Sensorimotor Performance; Behavioral Health Management; Attention Optimization; Stress Reduction; Fatigue Management; Cognitive Load; Environmental Modulations; Performance Enhancement; Non-Invasive Sensors; Adaptive Techology; Personalized Feedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Population (Experimental): With multiple testing periods per week over the course of 6 weeks. Participants will perform the standardized tasks both with and without deployment of the countermeasure during this period. Psychophysiological assessment and countermeasure deployment will be conducted with non-invasive sensors for physiological monitoring and non-invasive effectors.
  Interventions: Device: AttentivU

INTERVENTIONS:
Device: AttentivU — A device for continuous brain and physiology monitoring. It includes up to 8 EEG sensors as well as EOG and accelerometry which can be monitored in real-time for changes in attention, sleepiness, alertness, cognitive load, stress, and related psychological traits. The EEG data is analyzed in real-time to identify these states and this information can then be used to modulate "countermeasures" to the state--to either increase or decrease alertness or help counteract cognitive load sleepiness or stress conditions.

SUMMARY:
Crews of future long-duration exploration missions will have to cope with a wide range of stressors that present significant challenges for maintaining optimal performance. Crews will have to operate under conditions of high workload, reduced sleep and circadian dysregulation, limited sensory stimulation, confinement and extended separation from family and friends, and communication delays isolating them from real-time interaction with ground support, which may be particularly critical in the event of emergencies. These factors present significant risks to optimal cognitive/behavioral functioning and performance, across individuals and teams, and such challenges will only increase in criticality as human exploration moves beyond Earth's orbit to targets such as the Moon and Mars. To help mitigate these risks, Massachusetts General Hospital, along with collaborators at the Massachusetts Institute of Technology, will investigate a novel, personalized and scalable, closed-loop platform technology for on-board behavioral health management-one which adapts the local working environment to optimize performance based on biosensor feedback.

DETAILED DESCRIPTION:
1. Background and Significance

   Crews of future long-duration space exploration missions will have to cope with a wide range of stressors that present significant challenges for maintaining optimal performance. Crews will have to operate under conditions of high workload, reduced sleep and circadian dysregulation, limited sensory stimulation, confinement and extended separation from family and friends [5], and communication delays isolating them from real-time interaction with ground support, which may be particularly critical in the event of emergencies. These factors present significant risks to optimal cognitive/behavioral functioning and performance, across individuals and teams, and such challenges will only increase in criticality as human exploration moves beyond Earth's orbit to targets such as the Moon and Mars.

   To help mitigate these risks, Massachusetts General Hospital, along with collaborators at the Massachusetts Institute of Technology, will investigate a novel, personalized and scalable, closed-loop platform technology for on-board behavioral health management-one which adapts an individual's local working environment to optimize performance, based on biosensor feedback.

   Countermeasures (CMs) to Maintain/Improve Performance The premise of this proposed work is dynamically modifying an individual's local environment to help optimize performance. Since video displays require complex electronics which may not function in deep space, the investigators will study the following non-video countermeasures (CMs).

   Auditory Stimulation: Acoustic cues are common in biofeedback systems, with beeps and chimes often used to help trigger attentional redirection. Other sound cues-including natural sounds like flowing water, or even music-can also induce performance-beneficial physiological responses, including predictable changes in arousal-related measures such as heart rate and EDA. The underlying beat of music has been shown to alter arousal, with different modulations promoting relaxation or increased attention. Previous work also suggests that music may impact complex task performance (e.g., driving), and may alter student learning, through its mediating effects on arousal and alertness.

   Haptic Stimulation: Haptic feedback-via vibration, touch, or electrical stimulation-can be administered through individual or coordinated arrays of actuators. Prior research shows that the body location of a vibrotactile device can determine stimulation effectiveness, with the back, neck, and wrist/forearm areas presenting particularly sensitive sites for pressure and vibration-based alerting. Rhythm, roughness, intensity, and frequency can also be altered optimize vibrotactile display design. Such haptic cues have previously proven effective in redirecting attention to promote user engagement during a task, as well as improving coordinated motor performance (e.g., ambulation and postural sway).

   Light Stimulation: Lighting brightness, intensity, and color all impact information processing. The chronobiological influence of blue light as a circadian pacemaker, for example, has been well established. Increasing light brightness has been shown to promote alertness, and color can strongly influence alertness as well as mood / emotional processing, with certain colors (e.g., green) being useful in the modulation of autonomic arousal. The frequency of light flickering can also affect behavioral performance, with 40Hz light flickering supporting increased attention/arousal, and 10Hz flickering supporting reduced arousal.

   Knowledge Gaps: The above prior findings demonstrate that modulations of auditory, haptic, and light stimuli can each produce reliable changes in neurocognitive and psychological state (e.g., arousal, attention) related to performance. However, limited work has been done to establish a direct connection between environmental augmentations and performance changes, and the investigators are not aware of any studies specifically targeting operationally-relevant (i.e., complex task) behavioral performance.

   Purpose: The purpose of the study is to explore if the investigators can reliably detect, measure and provide feedback to users to optimize their cognitive states using wearable devices that measure their brain activity and other physiological signals, with the goal of improving behavioral task performance.

   Study endpoints: Change in the user's performance level (enhancements or decrements) while performing experimental tasks.

   Study Structure: These studies will be conducted at MIT-which is a subcontract under the MGH (=prime) award from NASA (prime PI=Dr. Gary Strangman)-by the MIT investigators, with design and analysis support from the MGH investigators. All data collected-in de-identified, coded form only-will be transmitted to Dr. Strangman at MGH (via secure transfer.partners.org) for additional analysis and to implement the required data sharing back to NASA. MGH personnel will not have access to the coding key.
2. Specific Aims and Objectives

The overall goal is to explore if one can (1) reliably measure physiological signals to detect person's cognitive states such as attention, fatigue, cognitive load and stress, and (2) provide the feedback to the user to help improve behavioral states, questionnaires, and/or users' overall performance.

The investigators will quantify performance changes associated with simple sensory manipulations in both cognitive tasks and tasks that are relevant to spaceflight operations. Tasks will include a battery of cognitive tests as well as tasks that are operationally-relevant to NASA. Environmental manipulations will seek to maintain optimal attention, engagement, cognitive load, and alertness, as assessed by psychophysiological signatures.

Aim 1: Assess behavioral changes associated with auditory-based manipulations. Aim 2: Assess behavioral changes associated with haptic-based manipulations. Aim 3: Assess behavioral changes associated with light-based manipulations.

Hypotheses: For each Aim, the investigators hypothesize that the P-POP system's personal environment modulations (e.g., sound, haptics, light) will generate significant improvements in individuals' cognitive and operational performance.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Must be between the ages of 18 to 64
* Normal or corrected-to-normal vision and hearing
* Ability to sit still and stay awake during the experimental sessions

Exclusion Criteria:

* Diagnosis with Neurological or psychiatric disorder
* Participation in a prior study associated with this protocol (due to the learning- curve on some of the behavioral tests)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
N-Back Task | 6 Weeks
  A cognitive assessment designed to measure working memory speed and accuracy. During the task, participants are presented with a sequence of stimuli (letters, numbers, or spatial locations) and must indicate whether the current stimulus matches the one presented earlier. Performance is assessed through reaction time, accuracy, and response variability, providing insight into both cognitive processing speed and working memory capacity.
Psychomotor Vigilance Test (PVT) | 6 Weeks
  A Validated neurobehavioral assessment of sustained attention and reaction time performance. The task measures the participant's ability to detect and respond to a visual stimulus, typically a randomly-timed cue presented on a screen. Key outcome measures include mean reaction time, lapses (responses exceeding a defined threshold, typically 500 ms), and false starts (premature responses).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MIT Media Lab, Cambridge, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts